CLINICAL TRIAL: NCT04897815
Title: Fasting and Postprandial Cerebral Blood Flow in Type 2 Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: LJB-01
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus; Cerebral Blood Flow
Keywords: Type 2 Diabetes Mellitus; Cerebral blood flow
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 20 patients with type 2 diabetes mellitus: Fasting blood glucose and TCD will be measured in 20 patients with type 2 diabetes mellitus, and the data of Vm, PI and cerebrovascular reactivity of cerebral artery will be obtained. One hour after drinking 300ml lukewarm water which has dissolved 75g glucose powder, the blood glucose will be detected again and TCD examination will be performed again.
- 20 healthy volunteers whose sex and age and BMI matched with the experimental group: Fasting blood glucose and TCD will be measured in healthy control group, and the data of Vm, PI and cerebrovascular reactivity of cerebral artery will be obtained. One hour after drinking 300ml lukewarm water which has dissolved 75g glucose powder, the blood glucose will be detected again and TCD examination will be performed again.

SUMMARY:
The purpose of this study is to explore the changes of fasting and postprandial cerebral blood flow in patients with type 2 diabetes mellitus. Some studies have proved that non-fasting blood glucose concentration is an independent predictor of ischemic stroke and lacunar infarction. At present, there are differences in cerebral blood flow velocity between diabetic patients and healthy controls. Therefore, it is of certain significance to explore the changes of fasting and postprandial cerebral blood flow in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
In China, due to the aging population and the increase in obesity, the incidence of diabetes is on the rise. Diabetes is the main independent risk factor for cerebrovascular diseases, especially ischemic stroke. Some studies have proved that non-fasting blood glucose concentration is an independent predictor of ischemic stroke and lacunar infarction. Transcranial Doppler (TCD) can evaluate intracranial blood flow patterns real-time and reliably, and provide information about cerebral hemodynamics, cerebrovascular reactivity and various pathological changes. At present, there are some differences in the study of cerebral blood flow velocity in diabetic patients. The purpose of our study is to determine the changes of cerebral blood flow on an empty stomach and 1 hour after meal in patients with type 2 diabetes. In this study, 20 patients with type 2 diabetes mellitus will be selected as the experimental group. 20 healthy volunteers whose sex and age and BMI matched with the experimental group will be selected as the control group. Fasting blood glucose and TCD will be measured in the two groups, and the data of mean flow velocity (Vm), Gosling's pulsatility index (PI) and cerebrovascular reactivity of cerebral artery will be obtained. One hour after drinking 300ml lukewarm water which has dissolved 75g glucose powder, the blood glucose will be detected again and TCD examination will be performed again. Finally, the data will be collected for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Trial group

  1. Study time: June 1, 2021, to January 1, 2022;
  2. Study site: The First Affiliated Hospital of Shandong First Medical University;
  3. 25-65 years old (including upper and lower limits), male or female;
  4. Meeting the diagnostic criteria of type 2 diabetes (according to 1997 WHO's diagnostic criteria for type 2 diabetes);
  5. Fasting blood glucose < 10 mmol/L;
  6. HbA1c ≤ 11.0%.
* Control group

  1. Study time: June 1, 2021, to January 1, 2022;
  2. Study site: The First Affiliated Hospital of Shandong First Medical University;
  3. Relatively healthy people without type 2 diabetes mellitus diagnosis;
  4. Participants whose sex and age and BMI matched with the experimental group.

Exclusion Criteria:

* Trial group and Control group

  1. Participants with diabetic retinopathy;
  2. Participants with diabetic neuropathy;
  3. Participants with diabetic nephropathy;
  4. Participants have unilateral or bilateral carotid plaque;
  5. Participants have a history of cardio-cerebrovascular disease;
  6. Participants have a history of respiratory disease;
  7. Participants complicated with hypertension;
  8. Participants complicated with hyperlipidemia;
  9. Participants have a smoking history (including previous smoking history);
  10. Participants complicated with malignant tumor.
  11. Participants are currently taking anticoagulants or vasodilators;
  12. Participants do not sign a written informed consent form.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes mellitus and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes of cerebral blood flow on fasting and 1 hour postprandial. | Data for each participant will be collected within 3 days.
  Detect changes in cerebral blood flow after fasting and 1 hour after meal by TCD, including changes in average cerebral blood flow velocity, PI, and cerebrovascular reactivity.

SECONDARY OUTCOMES:
The relationship between the fluctuation of blood glucose and the change of cerebral blood flow. | Data of all participants will be collected within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital